CLINICAL TRIAL: NCT04835376
Title: Percussion Palm Cup: Safety and Usability of Newly Designed Products in Infants and Children With Cystic Fibrosis
Brief Title: Percussion Palm Cup: Safety and Usability in Infants and Children With Cystic Fibrosis
Acronym: PPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Dina Brooks, Principal Investigator, West Park Healthcare Centre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 13112
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Cystic Fibrosis in Children
Keywords: Cystic Fibrosis; Chest Physiotherapy; Percussion Palm Cup; Children and Infants
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Randomized crossover intervention
Who Masked: Participant
Masking Description: The cups will be numbered, not identified by manufactured cup or 3D printed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Randomized Crossover: Percussion Palm Cup Safety and Usability - Cup 1 (Experimental): The standard percussor palm cups are made out of a soft vinyl material molded into shape. The outer diameter of the infant palm cup is 1-3/4 inches and there is a 1-inch diameter pocket inside this product similar to a suction cup.
  Interventions: Device: Percussion Palm Cup: Safety and Usability of Newly Designed Products in Infants and Children with Cystic Fibrosis
- Randomized Crossover: Percussion Palm Cup Safety and Usability - Cup 2 (Experimental): This product was developed by MMRI personnel using a small custom 3D printed plastic handle and a 0.93-inch, single bellow, Buna-N rubber suction cup. The handle was made on the MMRI's 3D printer using ABS plastic and the suction cup was sourced from McMaster Carr (#5427A106). The handle is made up of three pieces; top, base and a pin that is designed to fix the top, base and suction cup to each other. There is a small hole through the pin which helps relieve some of the pressure that builds in the suction cup during use. It is not shown in the image to the right, but the handle will be coated in Plasti Dip for added user comfort.
  Interventions: Device: Percussion Palm Cup: Safety and Usability of Newly Designed Products in Infants and Children with Cystic Fibrosis
- Randomized Crossover: Percussion Palm Cup Safety and Usability - Cup 3 (Experimental): This product was developed by MMRI personnel using a large custom 3D printed plastic handle and a 0.93-inch, single bellow, Buna-N rubber suction cup. The handle was made on the MMRI's 3D printer using ABS plastic and the suction cup was sourced from McMaster Carr (#5427A106). The handle is made up of three pieces; top, base and a pin that is designed to fix the top, base and suction cup to each other. There is a small hole through the pin which helps relieve some of the pressure that builds in the suction cup during use. It is not shown in the image to the right, but the handle will be coated in Plasti Dip for added user comfort.
  Interventions: Device: Percussion Palm Cup: Safety and Usability of Newly Designed Products in Infants and Children with Cystic Fibrosis

INTERVENTIONS:
Device: Percussion Palm Cup: Safety and Usability of Newly Designed Products in Infants and Children with Cystic Fibrosis — Patients/guardians/caregivers will be given 3 percussor palm cups to use over the course of 6 days. Each cup will be trialed for 2 days, allowing for equal time dedicated to each.

SUMMARY:
Cystic Fibrosis is the most prevalent fatal genetic disease affecting Canadian children and it primarily characterized by a thickening of pulmonary secretions and impaired mucociliary clearance. Chest physiotherapy has been widely used as a standard treatment for sputum mobilization and clearance for individuals with CF. Percussion is one such technique of chest physiotherapy for loosening trapped music within the lungs and can be completed manually or facilitated with a percussion cup. Unfortunately, the exclusive Canadian supplier for the widely use percussor cup has stopped distributing the cups, leaving many hospitals and therapy clinics searching for alternatives to continue airway clearance treatment. The goal of this project is to compare alternative palm cup solutions to the standard, and recommend safe alternative(s) that caregivers can have easy access to.

DETAILED DESCRIPTION:
An average adult hand may be too large and taxing for percussion on infants and children, therefore percussor palm cups facilitate caregivers and physiotherapists. The palm cup mimics the air compressed through cupped hands and can be used in conjunction with other physiotherapy techniques and has been shown to have a positive impact on symptoms. Engineers at McMaster University have developed 3D-printed prototypes to use with percussor cups that are made with material similar in consistency and flexibility to the no longer manufactured, standard cup. These cups will be tested in infants and children with cystic fibrosis recruited from the Cystic Fibrosis Clinic at McMaster Children's Hospital in Hamilton, Ontario.

Patients/guardians/caregivers will be given 3 percussor palm cups to use over the course of 6 days (one standard cup and two 3D-printed). Each cup will be trialed for 2 days, allowing for equal time dedicated to each. Demographic data and characteristics will be collected at baseline, and measures of safety and usability will be completed at the end of the week of use. Overall satisfaction will be recorded at the end of the questionnaire. Participants will be asked to rate percussion palm cups from least preferred to most preferred and an open-ended question to explain their reasoning on the experience.

Thus, the purpose of the study is to examine the safety, usability and user experience of newly designed percussion palm cups using 3-D printing. The results of this study will have important implication to the management of infants and children with CF given the percussion palm cup shortage.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children with CF under the age of 6 and their parent/guardian/caregiver to perform chest percussions using percussor palm cups.
* Participants must currently require regular chest physiotherapy.

Exclusion Criteria:

* A comorbid condition that is a contraindication for the use of percussor palm cups.
* Inability of parent/guardian/caregiver to complete written questionnaires due to visual or cognitive impairment.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Safety and user questionnaire | Through study completion, average 1 year
  Participants and families will be asked to report any adverse effects of the use of the PCC. These could include erythema of the skin, bruising or general discomfort using a 5-point Likert scale (1 = very disatisfied, 5 = very satisfied) and open-ended questions. A higher value on the Likert scale indicates a better outcome as the participant identifies that they were satisfied when using the cup. This will also be used to compare satisfaction between cups.
Usability using the Pictorial Single-Item Usability Scale (PSIUS) | Through study completion, average 1 year
  The Pictorial Single-Item Usability Scale (PSIUS) is an instrument used to measure perceived usability and satisfaction of each cup. This scale concludes three main visual elements that evaluate satisfaction and emotions experience while using a system or product. It uses visual images of disatisfaction to satisfaction, following a 9-point scale (-4 = very disatisfied, 4 = very satisfied). A higher number indicates a better experience when using the cup. This pictorial single-item scale will be used within our questionnaire to assess the overall rating of satisfaction and usability when using the Percussion Palm Cups.

SECONDARY OUTCOMES:
Quebec User Evaluation Utility Questionnaire (QUEST) | Through study completion, average 1 year
  The Quebec User Evaluation Utility Questionnaire (QUEST) is designed to evaluate user satisfaction and dissatisfaction with assistive devices. It is the most commonly used standardized instrument for measuring user satisfaction with a broad range of assistive technology devices. The revised QUEST 2.0 version includes a 12-item structure, with each item scored using a 5-point satisfaction scale (1= not satisfied at all, 5 = very satisfied). Additionally, the user is asked to comment on the source of their dissatisfaction or satisfaction on each item. We will use the applicable items (8 in total) Comfort, Dimensions, Simplicity of Use, Effectiveness, Durability, Adjustments, Safety, and Weight.
Overall satisfaction questionnaire | Through study completion, average 1 year
  Overall satisfaction and user experience will be recorded. Participants will be asked to discuss any concerns, discomfort when using the palm cup and rate percussion palm cups from least preferred to most preferred with open-ended questions to explain their reasoning with no minimum or maximum values. Each cup will be ranked as either first, second, and third choice (cup #1,2,3 = first, second or third choice in ranking). First choice indicates the best overall experience, last choice indicates the worst overall expereince or least preferred.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital Cystic Fibrosis Clinic, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Button BM, Heine RG, Catto-Smith AG, Olinsky A, Phelan PD, Ditchfield MR, Story I. Chest physiotherapy in infants with cystic fibrosis: to tip or not? A five-year study. Pediatr Pulmonol. 2003 Mar;35(3):208-13. doi: 10.1002/ppul.10227. PMID 12567389
- [Background] Flume PA, Robinson KA, O'Sullivan BP, Finder JD, Vender RL, Willey-Courand DB, White TB, Marshall BC; Clinical Practice Guidelines for Pulmonary Therapies Committee. Cystic fibrosis pulmonary guidelines: airway clearance therapies. Respir Care. 2009 Apr;54(4):522-37. PMID 19327189
- [Background] Riordan JR, Rommens JM, Kerem B, Alon N, Rozmahel R, Grzelczak Z, Zielenski J, Lok S, Plavsic N, Chou JL, et al. Identification of the cystic fibrosis gene: cloning and characterization of complementary DNA. Science. 1989 Sep 8;245(4922):1066-73. doi: 10.1126/science.2475911.
- [Background] Collins FS. Cystic fibrosis: molecular biology and therapeutic implications. Science. 1992 May 8;256(5058):774-9. doi: 10.1126/science.1375392.
- [Background] Gursli S, Sandvik L, Bakkeheim E, Skrede B, Stuge B. Evaluation of a novel technique in airway clearance therapy - Specific Cough Technique (SCT) in cystic fibrosis: A pilot study of a series of N-of-1 randomised controlled trials. SAGE Open Med. 2017 Mar 17;5:2050312117697505. doi: 10.1177/2050312117697505. eCollection 2017. PMID 28540046
- [Background] O'Sullivan BP, Freedman SD. Cystic fibrosis. Lancet. 2009 May 30;373(9678):1891-904. doi: 10.1016/S0140-6736(09)60327-5. Epub 2009 May 4. PMID 19403164
- [Background] Orenstein DM, Boat TF, Stern RC, Tucker AS, Charnock EL, Matthews LW, Doershuk CF. The effect of early diagnosis and treatment in cystic fibrosis: a seven-year study of 16 sibling pairs. Am J Dis Child. 1977 Sep;131(9):973-5. doi: 10.1001/archpedi.1977.02120220039005. PMID 900085
- [Background] Warnock L, Gates A. Chest physiotherapy compared to no chest physiotherapy for cystic fibrosis. Cochrane Database Syst Rev. 2015 Dec 21;2015(12):CD001401. doi: 10.1002/14651858.CD001401.pub3. PMID 26688006
- [Background] Punithavathi N, Ong LM, Irfhan Ali HA, Mohd Izmi IA, Dharminy T, Ang AH, Hadzlinda Z, Sivasangari S. A Pilot Randomized Control Cross over Study Evaluating the Effectiveness and Safety of Mechanical Percussor Compared with Conventional Chest Physiotherapy in Adults with Productive Cough. Med J Malaysia. 2014 Feb;69(1):16-20. PMID 24814623
- [Background] Blazey S, Jenkins S, Smith R. Rate and force of application of manual chest percussion by physiotherapists. Aust J Physiother. 1998;44(4):257-264. doi: 10.1016/s0004-9514(14)60385-8. PMID 11676741
- [Background] Gregson RK, Stocks J, Petley GW, Shannon H, Warner JO, Jagannathan R, Main E. Simultaneous measurement of force and respiratory profiles during chest physiotherapy in ventilated children. Physiol Meas. 2007 Sep;28(9):1017-28. doi: 10.1088/0967-3334/28/9/004. Epub 2007 Aug 21. PMID 17827650
- [Background] Hardy KA, Anderson BD. Noninvasive clearance of airway secretions. Respir Care Clin N Am. 1996 Jun;2(2):323-45. PMID 9390886
- [Background] Demers L, Weiss-Lambrou R, Ska B. Item analysis of the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST). Assist Technol. 2000;12(2):96-105. doi: 10.1080/10400435.2000.10132015. PMID 11508406
- [Background] Greulich T, Kehr K, Nell C, Koepke J, Haid D, Koehler U, Koehler K, Filipovic S, Kenn K, Vogelmeier C, Koczulla AR. A randomized clinical trial to assess the influence of a three months training program (gym-based individualized vs. calisthenics-based non-invidualized) in COPD-patients. Respir Res. 2014 Mar 25;15(1):36. doi: 10.1186/1465-9921-15-36. PMID 24666558
- [Background] Vaismoradi M, Turunen H, Bondas T. Content analysis and thematic analysis: Implications for conducting a qualitative descriptive study. Nurs Health Sci. 2013 Sep;15(3):398-405. doi: 10.1111/nhs.12048. Epub 2013 Mar 11. PMID 23480423